CLINICAL TRIAL: NCT02668861
Title: Influence of Oral Vitamin D3 on Wound Healing After Endonasal Endoscopic Sinus Surgery for Chronic Rhinosinusitis With Nasal Polyposis and Lower Vitamin D Levels
Brief Title: Effect of Oral Vitamin D3 on Chronic Rhinosinusitis Treatment in Adults With Lower Vitamin D Levels
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Jun Tian, Associate Professor, The First Affiliated Hospital of Shanxi Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FirstTianjunMU
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: interventions — Vitamin D; Budesonide

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Vitamin D+Budesonide Nasal Spray (Experimental): Vitamin D 4000IU/day for 8 weeks + Budesonide Nasal Spray 128ug/d for 8 week
  Interventions: Drug: Vitamin D; Drug: Budesonide Nasal Spray
- placebo+Budesonide Nasal Spray (Placebo Comparator): Placebo for 8 weeks + Budesonide Nasal Spray128ug/d for 8 week
  Interventions: Drug: Budesonide Nasal Spray; Other: placebo

INTERVENTIONS:
Drug: Vitamin D — Vitamin D 4000IU/day for 8 weeks
  Arms: Vitamin D+Budesonide Nasal Spray
Drug: Budesonide Nasal Spray — Budesonide Nasal Spray 128ug/d for 8 week
  Other Names: Rhinocort Aqua
Other: placebo — placebo for 8 weeks
  Arms: placebo+Budesonide Nasal Spray

SUMMARY:
The purpose of the study is to test the clinical efficacy of oral Vitamin D3 on Wound Healing in patients with Chronic Rhinosinusitis With Nasal Polyposis and Lower Vitamin D Levels After Endonasal Endoscopic Sinus Surgery

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinical diagnosis of Chronic Rhinosinusitis with nasal polyps 2. Be 18-60 years old of Chinese people and of either sex，the Han nationality 3. Vitamin D level of less than 30 ng/ml

Exclusion Criteria:

* 1. Women must not be pregnant, breast feeding 2. Chronic oral corticosteroid therapy 3. History of physician-diagnosed nephrolithiasis 4. Chronic diseases（ diabetes，Hypertension，renal insufficiency, severe liver disease） 5.prior surgeries of the paranasal sinuses 6. With an upper respiratory tract infection within 4 weeks of entering the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
VAS evaluation of usual symptoms in patients with CRSwNP | at 8 weeks after first drug intake
  The evaluated symptoms were nasal obstruction, anterior nasal discharge and post-nasal drip, smelling reduction and facial pain
Questionnaire：SNOT-20 evaluates the quality of Life | at 8 weeks after first drug intake
Change of Lund-Kennedy scores | at 8 weeks after first drug intake

SECONDARY OUTCOMES:
Inflammatory mediators in serum | 8 weeks
Histologic analysis of nasal mucosa | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Shanxi Medical University, Taiyuan, Shanxi, China